CLINICAL TRIAL: NCT02049957
Title: A Phase 1b/2 Study of Safety and Efficacy of MLN0128 (Dual TORC1/2 Inhibitor) in Combination With Exemestane or Fulvestrant Therapy in Postmenopausal Women With ER+/HER2- Advanced or Metastatic Breast Cancer That Has Progressed on Treatment With Everolimus in Combination With Exemestane or Fulvestrant
Brief Title: Safety and Efficacy Study of Sapanisertib in Combination With Exemestane or Fulvestrant in Postmenopausal Women With Estrogen Receptor Positive/Human Epidermal Growth Factor Receptor 2 Negative (ER+/HER2-) Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C31001; 2014-001921-34 (EudraCT Number); U1111-1195-3894 (Registry Identifier: WHO)
Record Dates: First submitted 2013-12-12; First posted 2014-01-30 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Sapanisertib; MLN0128
MeSH Terms: conditions — Breast Neoplasms | interventions — sapanisertib; Fulvestrant; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane (Experimental): Sapanisertib 5 mg, unmilled active pharmaceutical ingredient (API) capsule, once daily in a 28-day cycle plus exemestane 25 mg, tablets, once daily in a 28-day cycle (Up to 12 cycles).
  Interventions: Drug: Sapanisertib; Drug: Exemestane
- Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant (Experimental): Sapanisertib 5 mg, unmilled API capsule, once daily in a 28-day cycle plus fulvestrant 500 mg, injection, intramuscularly (IM), once on Day 1 of each cycle (Up to 57 cycles).
  Interventions: Drug: Sapanisertib; Drug: Fulvestrant
- Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane (Experimental): Sapanisertib 3 mg, milled API capsule, once daily in a 28-day cycle plus exemestane 25 mg, tablets, once daily in a 28-day cycle (Up to 8 cycles).
  Interventions: Drug: Sapanisertib; Drug: Exemestane
- Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant (Experimental): Sapanisertib 3 mg, milled API capsule, once daily in a 28-day cycle up to 14 cycles plus fulvestrant 500 mg, injection, IM, once on Day 1 of each cycle (Up to 14 cycles).
  Interventions: Drug: Sapanisertib; Drug: Fulvestrant
- Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane (Experimental): Sapanisertib 4 mg, milled API capsule, once daily, in a 28-day cycle plus exemestane 25 mg, tablets, once daily in a 28-day cycle (Up to 18 cycles).
  Interventions: Drug: Sapanisertib; Drug: Exemestane
- Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) (Experimental): Sapanisertib 4 mg, milled API capsule once daily in a 28-day cycle plus exemestane 25 mg, tablets, once daily in a 28-day cycle (Up to 14 cycles) in everolimus sensitive participants.
  Interventions: Drug: Sapanisertib; Drug: Exemestane
- Phase 2:Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) (Experimental): Sapanisertib 4 mg, milled API capsule once daily in a 28-day cycle plus fulvestrant 500 mg, injection IM, once on Day 1 of each cycle (Up to 17 cycles) in everolimus sensitive participants.
  Interventions: Drug: Sapanisertib; Drug: Fulvestrant
- Phase 2: Sapanisertib 4 mg+Exemestane (Everolimus Resistant) (Experimental): Sapanisertib 4 mg, milled API capsule, once daily, in a 28-day cycle plus once daily in a 28-day cycle (Up to 12 cycles) in everolimus resistant participants.
  Interventions: Drug: Sapanisertib; Drug: Exemestane
- Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant) (Experimental): Sapanisertib 4 mg, milled API capsule, once daily in a 28-day cycle plus fulvestrant 500 mg, injection IM, once on Day 1 of each cycle (Up to 9 cycles) in everolimus resistant participants.
  Interventions: Drug: Sapanisertib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Sapanisertib — Sapnisertib capsules
  Other Names: MLN0128
Drug: Fulvestrant — Fulvestrant IM injection.
  Arms: Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant; Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant; Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant); Phase 2:Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive)
Drug: Exemestane — Exemestane tablets.
  Arms: Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane; Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane; Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane; Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive); Phase 2: Sapanisertib 4 mg+Exemestane (Everolimus Resistant)

SUMMARY:
This is a phase 1b/2 study of the safety and efficacy of sapanisertib (MLN0128) in combination with exemestane or fulvestrant therapy in women with estrogen receptor positive/human epidermal growth factor receptor 2 negative (ER+/HER2-) advanced or metastatic breast cancer who progressed on treatment with everolimus in combination with exemestane or fulvestrant.

DETAILED DESCRIPTION:
The drug being tested in this study is called sapanisertib (MLN0128). Sapanisertib is being tested in women with estrogen receptor positive/human epidermal growth factor receptor 2 negative (ER+/HER2-) advanced or metastatic breast cancer who progressed on treatment with everolimus. This study will look at the safety and efficacy of sapanisertib when given in combination with exemestane or fulvestrant.

The study enrolled 118 patients. This study has two phases: phase 1 and phase 2. Phase 1 has 2 parts. In part 1 of phase 1, unmilled active pharmaceutical ingredient (API) capsules were administered, while in part 2, capsules based on milled API were administered.

* Phase 1 (Part 1): sapanisertib 5 mg (unmilled) + exemestane
* Phase 1 (Part 1): sapanisertib 5 mg (unmilled) + fulvestrant
* Phase 1 (Part 2): sapanisertib 3 mg (milled) + exemestane
* Phase 1 (Part 2): sapanisertib 3 mg (milled) + fulvestrant
* Phase 1 (Part 2): sapanisertib 4 mg (milled) + exemestane

In phase 2, participants were enrolled into one of 2 parallel cohorts, depending on the quality and/or duration of their prior response to everolimus in combination with either exemestane (any country) or fulvestrant (US only).

Everolimus-Resistant Cohort: patients who had progressed on treatment with everolimus in combination with either exemestane (any country) or fulvestrant (US only) without achieving an objective response (CR or PR) or after achieving stable disease for <6 months as their best response.

Everolimus-Sensitive Cohort: participants who had progressed on treatment after achieving a CR or PR of any duration, or stable disease for ≥6 months with prior everolimus treatment in combination with either exemestane (any country) or fulvestrant (US only). Participants were to receive MLN0128 in combination with the same dose of the previously administered treatment (exemestane [any country] or fulvestrant [US only]).

This multi-center trial will be conducted worldwide. The overall time to participate in this study was 52 months. Participants made multiple visits to the clinic and were contacted by telephone every 3 months for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

Phase 1b and Phase 2

1. Advanced or metastatic breast cancer.
2. Histological or cytological confirmation of ER+ status (defined as > 1% positive tumor cells), and histological or cytological confirmation of HER2-negative (HER2-) status by local laboratory testing using criteria in the American Society of Oncology (ASCO)/College of American Pathologists (CAP) Clinical Practice Guideline update.
3. Female patients 18 years of age or older who are postmenopausal for at least 1 year before the Screening visit, where menopause is defined by: Age ≥ 55 years and 1 year or more of amenorrhea. Surgical menopause with bilateral oophorectomy

   Age < 55 years and 1 year or more of amenorrhea, with an estradiol assay < 20 pg/mL

   Note: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression.
4. Have a history of brain metastasis are eligible for the study provided that all the following criteria are met:

   Brain metastases which have been treated
   * No evidence of disease progression for ≥ 3 months or hemorrhage after treatment
   * Off-treatment with dexamethasone for 4 weeks before administration of the first dose of MLN0128
   * No ongoing requirement for dexamethasone or anti-epileptic drugs
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
6. Clinical laboratory values as specified below within 4 weeks before the first dose of MLN0128:

   * Bone marrow reserve consistent with absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; platelet count ≥ 100 x 10^9/L; hemoglobin ≥ 9 g/dL
   * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present)
   * Creatinine clearance ≥ 50 mL/min based either on Cockcroft-Gault estimate or based on a 12- or 24-hour urine collection
   * Fasting serum glucose ≤ 130 mg/dL and fasting triglycerides ≤ 300 mg/dL
7. Left ventricular ejection fraction (LVEF) within 5 absolute percentage points of institutional standard of normal as measured by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) within 4 weeks before the first dose of MLN0128 (ie, if the institutional standard of normal is 50%, LVEF may be as low as 45% to be eligible for the study).
8. Able to provide paraffin blocks or a minimum of 10 unstained slides of available archival tumor tissues (paraffin blocks are preferred). If archival tumor tissue is not available, a tumor biopsy may be performed before the patient begins treatment with MLN0128. If fewer than 10 slides are available or the tumor content/area requirements are not met, study eligibility will be determined upon discussion with the sponsor.
9. Ability to swallow oral medications, willingness to perform mucositis prophylaxis, and suitable venous access for the study-required blood sampling.
10. Voluntary written consent must be given before the performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

    Phase 1b Only: In addition to the previously mentioned inclusion criteria, each patient must meet the following inclusion criterion to be enrolled in the phase 1b portion of the study:
11. Patients may have SD or disease progression during their most recent treatment with exemestane or fulvestrant, or everolimus in combination with either exemestane (any country) or fulvestrant (US only). Exemestane or fulvestrant in combination with MLN0128 can also be initiated as a new line of therapy.

    Phase 2 Only: In addition to the previously mentioned inclusion criteria, each patient must meet all of the following inclusion criteria to be enrolled in the phase 2 portion of the study:
12. Measurable disease defined as follows:

    * At least 1 extra-osseous lesion that can be accurately measured in at least 1 dimension. The lesion must measure ≥ 20 mm with conventional imaging techniques or ≥ 10 mm with spiral computed tomography (CT) or magnetic resonance imaging (MRI), or
    * Bone lesions (lytic or mixed [lytic plus sclerotic]) in the absence of measurable disease as defined above
13. Patients must have had disease progression during treatment with everolimus in combination with either exemestane (any country) or fulvestrant (US only) (duration of treatment ≥ 4 weeks) and must have tolerated everolimus treatment in combination with exemestane (any country) or fulvestrant (US only) adequately according to the treating physician's judgment. Everolimus in combination with exemestane or fulvestrant is not required to be the most recent treatment before enrollment, but progression on the most recent anticancer therapy is required for enrollment.

Exclusion Criteria

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

Phase 1b and Phase 2

1. Prior anticancer therapy or other investigational therapy within 2 weeks before administration of the first dose of MLN0128 (except for exemestane or fulvestrant, which should be continued). Treatment with everolimus must be discontinued 2 weeks before administration of the first dose of MLN0128.
2. Chronic concomitant therapy with bisphosphonates or denosumab for the prevention of bone metastases. Concomitant treatment with bisphosphonates or denosumab is permitted for treatment of osteoporosis or management of existing bone metastases if initiated at least 4 weeks before administration of the first dose of MLN0128.
3. Initiation of treatment with hematopoietic growth factors, transfusions of blood and blood products, or systemic corticosteroids (either IV or oral steroids, excluding inhalers) within 1 week before administration of the first dose of MLN0128 (patients already receiving erythropoietin on a chronic basis for ≥ 4 weeks are eligible).
4. Previous treatment with dual PI3K/mTOR inhibitors or TORC1/2 inhibitors.
5. Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of MLN0128.
6. Poorly controlled diabetes mellitus defined as glycosylated hemoglobin (HbA1c) > 7%; patients with a history of transient glucose intolerance due to corticosteroid administration may be enrolled in this study if all other inclusion/exclusion criteria are met.
7. Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise participation of the patient in the study.
8. Known human immunodeficiency virus infection.
9. History of any of the following within the last 6 months before administration of the first dose of MLN0128:

   * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
   * Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures
   * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation, or ventricular tachycardia)
   * Placement of a pacemaker for control of rhythm
   * New York Heart Association Class III or IV heart failure
   * Pulmonary embolism
10. Significant active cardiovascular or pulmonary disease before administration of the first dose of MLN0128, including:

    * Uncontrolled hypertension (ie, systolic blood pressure > 180 mm Hg; diastolic blood pressure > 95 mm Hg)
    * Pulmonary hypertension
    * Uncontrolled asthma or oxygen saturation < 90% by arterial blood gas analysis or pulse oximetry on room air
    * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention; or history of valve replacement
    * Medically significant (symptomatic) bradycardia
    * History of arrhythmia requiring an implantable cardiac defibrillator
    * Baseline prolongation of the rate-corrected QT interval (QTc; eg, repeated demonstration of QTc interval > 480 ms, or history of congenital long QT syndrome, or torsades de pointes)
11. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of MLN0128 or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

    Phase 1b Only: In addition to the previously mentioned exclusion criteria, patients meeting the following exclusion criterion are not to be enrolled in the phase 1b portion of the study:
12. More than 3 prior chemotherapy regimens for locally advanced or metastatic disease.

    Phase 2 Only: In addition to the previously mentioned exclusion criteria, patients meeting the following exclusion criterion are not to be enrolled in the phase 2 portion of the study:
13. More than 1 prior chemotherapy regimen for locally advanced or metastatic disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal Women With ER/PR+ Metastatic Breast Cancer.
Enrollment: 118 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (40):
- United States (30):
  - Los Angeles Hematology, Los Angeles, California
  - University of California at San Francisco (PARENT), San Francisco, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lakewood, Colorado
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - University of Kansas Medical Center Research Institute, Inc., Westwood, Kansas
  - Holy Cross Hospital, Silver Spring, Maryland
  - Henry Ford Medical Center, Novi, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Weill Cornell Medical College New York Presbyterian Hospital, New York, New York
  - Eastchester Center for Cancer Care / BRANY, The Bronx, New York
  - University of Cincinnati Physicians Company, LLC, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Texas Oncology, P.A. - Beaumont, Beaumont, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Millennium Oncology, Houston, Texas
  - Texas Health Physicians Group, Plano, Texas
  - Cancer Care Network of South Texas - SAT&BC, San Antonio, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Virginia Oncology Associates - Hampton, Chesapeake, Virginia
  - Oncology and Hematology Assoc. of SW VA, Inc., Salem, Virginia
  - West Virginia University, Morgantown, West Virginia
- Belgium (6):
  - UZ Antwerpen, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - GHdC Notre Dame, Charleroi
  - Centre Hospitalier de l'Ardenne, Libramont
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Wilrijk
- France (4):
  - Centre Francois Baclesse, Caen, Calvados
  - Centre Catherine de Sienne, Nantes, Loire Atlantique
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Sarthe
  - Institut Sainte Catherine, Avignon, Vaculuse

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Lim B, Potter DA, Salkeni MA, Silverman P, Haddad TC, Forget F, Awada A, Canon JL, Danso M, Lortholary A, Bourgeois H, Tan-Chiu E, Vincent S, Bahamon B, Galinsky KJ, Patel C, Neuwirth R, Leonard EJ, Diamond JR. Sapanisertib Plus Exemestane or Fulvestrant in Women with Hormone Receptor-Positive/HER2-Negative Advanced or Metastatic Breast Cancer. Clin Cancer Res. 2021 Jun 15;27(12):3329-3338. doi: 10.1158/1078-0432.CCR-20-4131. Epub 2021 Apr 5. PMID 33820779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 40 investigative sites in Belgium, France and the United States from 13 February 2014 to 03 July 2018.
Pre-assignment Details: Postmenopausal women with estrogen receptor positive/human epidermal growth factor receptor-2 negative advanced/metastatic breast cancer who progressed with everolimus (everolimus sensitive-achieved CR/PR of any duration/stable disease for ≥6 months; resistant-without CR/PR/SD < 6 months) were enrolled to receive MLN0128+exemestane/fulvestrant.
Groups:
- Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive): Sapanisertib 4 mg, milled API capsule once daily in a 28-day cycle plus fulvestrant 500 mg, injection IM, once on Day 1 of each cycle (Up to 17 cycles) in everolimus sensitive participants.
- Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant): Sapanisertib 4 mg, milled API capsule, once daily, in a 28-day cycle plus exemestane 25 mg, tablets, once daily in a 28-day cycle (Up to 12 cycles) in everolimus resistant participants.
Period: Overall Study
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant)
Started | 6 | 6 | 3 | 3 | 6 | 43 | 8 | 35 | 8
Completed (Completed=Completed Study Treatment) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 3 | 3 | 6 | 43 | 8 | 35 | 8
Not completed — Progressive Disease | 5 | 4 | 2 | 2 | 6 | 35 | 7 | 26 | 6
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 5 | 0 | 6 | 1
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population was defined as all participants who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant) | Total
Number analyzed (Participants) | 6 | 6 | 3 | 3 | 6 | 43 | 8 | 35 | 8 | 118
Age, Continuous [Mean (Full Range); unit: years] | 61.3 [52 to 74] | 56.2 [42 to 67] | 54.0 [39 to 62] | 52.3 [48 to 56] | 59.5 [33 to 75] | 58.9 [37 to 83] | 52.1 [32 to 73] | 58.8 [33 to 74] | 58.5 [47 to 70] | 57.31 [32 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 3 | 6 | 43 | 8 | 35 | 8 | 118
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 6 | 6 | 3 | 3 | 5 | 36 | 8 | 29 | 7 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 6 | 1 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 5 | 2 | 2 | 6 | 36 | 8 | 25 | 8 | 98
  Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 6
  Black or African American | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 1 | 0 | 7
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 4
  Other | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 3 | 3 | 6 | 30 | 8 | 25 | 8 | 95
  Belgium | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 7 | 0 | 16
  France | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 0 | 7
Height [Mean (Full Range); unit: cm] — Population: Number analyzed is the number of participants with data available for height.
  cm
    number analyzed (Participants) | 6 | 6 | 3 | 3 | 6 | 42 | 8 | 33 | 7 | 114
    (all) | 167.1 [160 to 177] | 165.7 [159 to 175] | 167.0 [160 to 175] | 170.8 [166.4 to 176] | 161.1 [155 to 165] | 163.5 [152 to 179] | 165.7 [158 to 175] | 164.5 [150 to 183] | 163.7 [154 to 177] | 165.02 [150 to 183]
Weight [Mean (Full Range); unit: kg] — Population: Number analyzed is the number of participants with data available for weight.
  kg
    number analyzed (Participants) | 6 | 6 | 3 | 3 | 6 | 43 | 8 | 34 | 8 | 117
    (all) | 69.18 [52.0 to 93.0] | 69.45 [52.6 to 120.2] | 70.57 [57.2 to 77.7] | 64.34 [59.5 to 69.4] | 63.63 [54.9 to 77.1] | 72.10 [47.2 to 123.7] | 67.45 [46.5 to 90.5] | 71.60 [50.0 to 114.0] | 82.10 [49.8 to 139.0] | 70.37 [46.5 to 139]

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. This includes any newly occurring event, or a previous condition that has increased in severity or frequency since the administration of study drug.
  A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event. Relationship of each AE to study drug will be determined by the Investigator.
Time Frame: First dose of study drug through 30 days after the last dose (Up to 52 months)
Population: Safety Population included participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane
Number analyzed (Participants) | 6 | 6 | 3 | 3 | 6
Participants
  Any AE | 6 | 6 | 3 | 3 | 6
  SAEs | 1 | 2 | 0 | 0 | 2

2. Primary Outcome: Phase 2: Clinical Benefit Rate at 16 Weeks (CBR-16)
Description: CBR-16 was defined as the percentage of participants who achieved confirmed complete response (CR) or partial response (PR) of any duration or had confirmed stable disease (SD) as best response and the first 2 or more post baseline scans had PR/SD and the duration of SD was >112 days. Disease response was assessed for target lesions by computed tomography (CT) or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines. CR is disappearance of all target lesions. PR is >=30% decrease in the sum of the longest diameter of target lesions. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression (PD).
Time Frame: Week 16
Population: Response-Evaluable Population included participants who received at least 1 dose of study drug and had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant)
Number analyzed (Participants) | 43 | 8 | 35 | 8
percentage of participants | 44 [29.1 to 60.1] | 50 [15.7 to 84.3] | 23 [10.4 to 40.1] | 25 [3.2 to 65.1]

3. Secondary Outcome: Phase 2: Clinical Benefit Rate at 24 Weeks (CBR-24)
Description: CBR-24 was defined as the percentage of participants who achieved confirmed CR or PR at any time or had confirmed SD as best response and the first 2 or more post baseline scans had PR/SD and the duration of stable disease was >168 days. Disease response was assessed for target lesions by CT or MRI according to RECIST version 1.1 guidelines. CR is disappearance of all target lesions. PR is >=30% decrease in the sum of the longest diameter of target lesions. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant)
Number analyzed (Participants) | 43 | 8 | 35 | 8
percentage of participants | 28 [15.3 to 43.7] | 38 [8.5 to 75.5] | 23 [10.4 to 40.1] | 25 [3.2 to 65.1]

4. Secondary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with confirmed CR or PR as per RECIST version1.1 guidelines. CR is disappearance of all target lesions. PR is >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Baseline then every 2 cycles from Cycles 2 through 6, and every 3 cycles thereafter in a 28-day cycle up to End of Treatment (EOT) (Up to 24 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant)
Number analyzed (Participants) | 43 | 8 | 35 | 8
percentage of participants | 7 [1.5 to 19.1] | 13 [1 to 52.7] | 0 [0 to 0] | 13 [1 to 52.7]

5. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: PFS is defined as the time in months from the date of first dose of study treatment to the date of the first documented disease progression or death. Disease progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 mm in the sum of diameters of target lesions; or the appearance of one or more new lesions.
Time Frame: Baseline then every 2 cycles from Cycles 2 through 6, and every 3 cycles thereafter in a 28-day cycle, then every 3 months after EOT until disease progression or death (Up to 24 months)
Population: Safety Population included participants who received at least 1 dose of study drug. For a participant whose disease had not progressed and was last known to be alive, PFS was censored at the last response assessment that was stable disease or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant)
Number analyzed (Participants) | 43 | 8 | 35 | 8
months | 4.1 [1.9 to 5.5] | 5.5 [1.8 to NA] — Upper limit of Confidence Interval (CI) was not reached due to low number of participants with events. | 3.3 [1.9 to 3.7] | 5.4 [1.7 to 8.3]

6. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is the time in months from start of study treatment to date of death due to any cause. Data for the analysis of OS included the censored data at the timepoint that the participant was last known to be alive.
Time Frame: Up to 24 months
Population: Safety Population included participants who received at least 1 dose of study drug. Participants without documentation of death at the time of analysis were censored at the date last known to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant)
Number analyzed (Participants) | 43 | 8 | 35 | 8
months | 15.9 [14.1 to 19.5] | 20.7 [8.6 to 20.7] | 14.0 [10.6 to 16.0] | 13.0 [4.1 to 21.3]

7. Secondary Outcome: Phase 2: Best Percent Change From Baseline in Tumor Size
Time Frame: Baseline to Month 24
Population: Participants from Safety Population included participants who received at least 1 dose of study drug and provided both baseline and at least one post-baseline disease response.
Measure: Mean (Standard Deviation); unit: percentage change in tumor size
Arm/Group | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant)
Number analyzed (Participants) | 36 | 7 | 27 | 7
percentage change in tumor size | -0.46 (34.89) | 0.96 (38.98) | 1.76 (31.14) | -18.91 (19.71)

8. Secondary Outcome: Phase1: Cmax: Maximum Observed Plasma Concentration for Sapanisertib
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1 pre-dose and multiple timepoints (Up to 8 hours) post-dose
Population: Pharmacokinetic (PK) Population included participants with sufficient dosing and PK data to reliably estimate PK parameters. PK data was not available for Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant arm group at Cycle 1 Day 15. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane
Number analyzed (Participants) | 6 | 5 | 3 | 3 | 6
ng/mL
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 0 | 3 | 2 | 6
  Cycle 1 Day 15 | 57.72 (9.927) |  | 47.40 (6.583) | 50.90 (23.476) | 45.37 (9.644)
  Cycle 2 Day 1: number analyzed (Participants) | 5 | 5 | 3 | 3 | 5
  Cycle 2 Day 1 | 38.68 (20.551) | 44.96 (34.459) | 43.47 (0.874) | 45.30 (16.235) | 44.68 (8.636)

9. Secondary Outcome: Phase 1: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Sapanisertib
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1 pre-dose and multiple timepoints (Up to 8 hours) post-dose
Population: PK Population included participants with sufficient dosing and PK data to reliably estimate PK parameters. PK data was not available for Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant arm group at Cycle 1 Day 15. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane
Number analyzed (Participants) | 6 | 5 | 3 | 3 | 6
hour
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 0 | 3 | 2 | 6
  Cycle 1 Day 15 | 3.005 [0.58 to 7.30] |  | 0.600 [0.45 to 1.00] | 1.035 [1.00 to 1.07] | 2.000 [0.50 to 3.55]
  Cycle 2 Day 1: number analyzed (Participants) | 5 | 5 | 3 | 3 | 5
  Cycle 2 Day 1 | 2.280 [0.85 to 3.58] | 3.500 [0.92 to 4.03] | 0.980 [0.68 to 1.00] | 1.000 [0.48 to 1.12] | 2.000 [0.50 to 3.77]

10. Secondary Outcome: Phase 1: AUC(0-24): Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours for Sapanisertib
Description: AUC(0-24) is the area under the plasma concentration-time curve of the samples collected up to 8 hours and extrapolated up to 24 hours.
Time Frame: Cycle 1 Day 15 pre-dose and multiple timepoints (Up to 8 hours) post-dose, extrapolated to 24 hours post-dose
Population: Participants from PK Population included participants with sufficient dosing and PK data to reliably estimate PK parameters. PK data was not available for Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant arm group at Cycle 1 Day 15. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane
Number analyzed (Participants) | 6 | 0 | 3 | 2 | 5
h*ng/mL | 577.081 (331.9813) |  | 178.063 (46.1416) | 332.618 (228.5641) | 277.626 (64.0661)

11. Secondary Outcome: Phase 1: AUC(0-last): Area Under the Plasma Concentration-time Curve From Time 0 to Last Extrapolated Concentration Over the Dosing Interval for Sapanisertib
Description: AUC(0-last) is the area under the plasma concentration-time curve of the samples collected up to 8 hours and extrapolated up to last time point.
Time Frame: Cycle 1 Day 15 pre-dose and multiple timepoints (Up to 8 hours) post-dose, extrapolated to last timepoint
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane
Number analyzed (Participants) | 6 | 5 | 3 | 3 | 6
h*ng/mL
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 0 | 3 | 2 | 6
  Cycle 1 Day 15 | 577.081 (331.9813) |  | 164.123 (52.6287) | 332.618 (228.5641) | 251.165 (83.7121)
  Cycle 1 Day 2: number analyzed (Participants) | 5 | 5 | 3 | 3 | 5
  Cycle 1 Day 2 | 101.599 (51.0248) | 109.496 (82.3968) | 89.576 (15.0117) | 109.548 (52.8500) | 116.557 (8.6059)

12. Secondary Outcome: Phase 1: Terminal Elimination Half-life (T1/2) for Sapanisertib
Time Frame: Cycle 1 Day 15 pre-dose and multiple timepoints (Up to 8 hours) post-dose
Population: Participants from PK Population, participants with sufficient dosing and PK data to reliably estimate PK parameters. PK data was not available for Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant arm group at Cycle 1 Day 15.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane
Number analyzed (Participants) | 2 | 0 | 3 | 2 | 4
hour | 6.639 (1.2176) |  | 3.161 (1.6585) | 7.777 (2.9177) | 5.370 (1.4638)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose (Up to 52 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/3 | 0/3 | 1/6 | 0/43 | 0/35 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 0/3 | 0/3 | 2/6 | 11/43 | 5/35 | 3/8 | 2/8
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/3 | 3/3 | 6/6 | 43/43 | 35/35 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane (N=6) | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant (N=6) | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane (N=3) | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant (N=3) | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane (N=6) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) (N=43) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) (N=35) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) (N=8) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant) (N=8)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with Sapanisertib 4 mg+Exemestane and was not related
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Part 1): Sapanisertib 5 mg + Exemestane (N=6) | Phase 1 (Part 1): Sapanisertib 5 mg + Fulvestrant (N=6) | Phase 1 (Part 2): Sapanisertib 3 mg + Exemestane (N=3) | Phase 1 (Part 2): Sapanisertib 3 mg + Fulvestrant (N=3) | Phase 1 (Part 2): Sapanisertib 4 mg + Exemestane (N=6) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Sensitive) (N=43) | Phase 2: Sapanisertib 4 mg + Exemestane (Everolimus Resistant) (N=35) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Sensitive) (N=8) | Phase 2: Sapanisertib 4 mg+Fulvestrant (Everolimus Resistant) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 6 | 6 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thyroid disorder (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal scar (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 2 | 2 | 4 | 17 | 9 | 3 | 6
Nausea (Gastrointestinal disorders) | 6 | 4 | 1 | 2 | 3 | 23 | 15 | 7 | 4
Stomatitis (Gastrointestinal disorders) | 5 | 3 | 0 | 0 | 2 | 10 | 8 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 3 | 10 | 10 | 1 | 5
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 6 | 5 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 5 | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 0 | 4 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 6 | 1 | 3 | 4 | 19 | 16 | 6 | 2
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 0 | 3 | 3 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 7 | 5 | 3 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sphingomonas paucimobilis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 2 | 0 | 1 | 3 | 6 | 4 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 6 | 5 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 3 | 6 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 2
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Amylase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Protein urine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 1 | 1 | 1 | 16 | 9 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 0 | 0 | 1 | 11 | 16 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 3 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 7 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 0 | 3 | 2 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 2
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 8 | 4 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 7 | 3 | 2 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 11 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 5 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serotonin syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglossal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis in device (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucinations, mixed (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 1 | 8 | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 7 | 4 | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 3 | 3 | 11 | 6 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2 | 5 | 3 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 1 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT02049957/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT02049957/SAP_001.pdf